CLINICAL TRIAL: NCT02170480
Title: Does Pin Size Influence the Incidence of Knee Pain in Patients Undergoing Temporary Skeletal Traction?
Brief Title: Pin Size Influence the Incidence of Knee Pain
Status: Terminated | Type: Observational
Why Stopped: PI is moving to another university; resident researcher does not wish to continue study with another PI.
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 57624
Record Dates: First submitted 2014-06-18; First posted 2014-06-23 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2016-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It has been the investigators observation that large diameter traction pins cause more postoperative knee pain than smaller traction pins. To the investigators knowledge, no study to date has identified knee pain as a consequence of traction pin placement. Furthermore, no study has identified whether pin size has an effect on the incidence of postoperative knee pain. The goal of the present study is to establish whether use of temporary skeletal traction is associated with subsequent knee pain and to determine whether traction pin size influences the incidence and/or magnitude of knee pain.

Objective #1:

Determine whether pin size influences the incidence and/or severity of postoperative knee pain in patients who undergo temporary skeletal traction.

Hypothesis:

Larger traction pins are associated with an increase in both the incidence and severity of postoperative knee pain.

Objective#2:

Determine whether pin size affects musculoskeletal function in the postoperative period.

Hypothesis:

There is no difference between small and large traction pins in postoperative musculoskeletal function.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults
* At least 18 years old
* Injury (Pelvic, acetabular, or femoral fracture) requiring temporary skeletal traction.

Exclusion Criteria:

* Neurovascular compromise.
* Ipsilateral fractures presenting contraindication to skeletal traction
* Patients who are non-ambulatory.
* Patients less than 18 years of age.
* Patients who do not speak English.
* Ipsilateral ligamentous knee injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the University of Utah Trauma and/or Orthopaedic Trauma services indicated for skeletal traction pin placement based on the presence of a femoral diaphyseal fracture and/or certain pelvic and acetabular fractures.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
2000 IKDC Subjective Knee Evaluation form, and pin site Visual Analog Pain Scale (VAS) | Post-operative follow-up visits up to 1 year
  Questionaires to assess knee pain

SECONDARY OUTCOMES:
Short Musculoskeletal Function Questionnaire (SMFA) | Post-operative follow-up visits up to 1 year
  Questionaire to assess musculoskeletal function

CONTACTS AND LOCATIONS:
Overall Officials: Erik Kubiak, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States